CLINICAL TRIAL: NCT07052396
Title: A Prospective, Non-interventional, Multicenter Observational Study to Evaluate Long-term Effectiveness and Safety, Patient Characteristics and Subjective Patient-reported Outcomes of Dupilumab in Patients With COPD Under Real-world Conditions
Brief Title: Study to Evaluate Long-term Effectiveness and Safety, Patient Characteristics and Subjective Patient-reported Outcomes of Dupilumab in Patients With Chronic Obstructive Pulmonary Disease (COPD) Under Real-world Conditions
Acronym: ANEMO
Status: Recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS18596; U1111-1314-5561 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — dupilumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

INTERVENTIONS:
Drug: Dupilumab — This study will not administer any treatment, only observe the treatment as prescribed in real world clinical practice.

SUMMARY:
Study to evaluate the change of health-related quality of life, patient characteristics, efficacy and safety in Chronic Obstructive Pulmonary Disease (COPD) patients with Dupilumab therapy in a real-world setting over 24 months.

DETAILED DESCRIPTION:
Non-interventional Study. Patients receive Dupilumab in accordance with the summary of product characteristics in a real-world setting. The Dupilumab initiation must be independent of the study recruitment and patient data is documented based on clinical routine.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing and able to sign informed consent for use of their pseudonymized clinical data within the present non-intervention study.
* Adult participants.
* Participants with uncontrolled Chronic Obstructive Pulmonary Disease (COPD) despite long-acting muscarinic antagonist (LAMA)/ long-acting beta2-agonist (LABA)/ Inhaled Corticosteroid (ICS) (or LAMA/LABA if ICS are not appropriate) therapy and elevated blood eosinophils
* Participants newly initiated on dupilumab treatment as indicated in the dupilumab Summary of Product Characteristics (SmPC) in the specified label for COPD, determined by the treating physician, and independent of participation in the non-interventional study (NIS).

Exclusion Criteria:

* Participants not eligible for dupilumab treatment according to SmPC.
* Participation in an ongoing interventional or observational study or participation in an interventional or observational study up to 12 months before enrolment that might, in the treating physician's opinion, influence the assessments for the current study.
* Any acute or chronic condition that, in the treating physician´s opinion, would limit the participants´s ability to complete questionnaires or to participate in this study or impact the interpretation of the results.
* Participants hospitalized due to an exacerbation of their COPD within the last 4 weeks prior to enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be screened, enrolled, and documented by their treating physician. To avoid any selection bias, all eligible participants will be invited to participate in this study in the order in which their eligibility is determined (consecutive recruitment). Participants will be treated within clinical routine practice and according to the current standard of care. Participants who permanently discontinue dupilumab treatment and therefore terminate the study prior to the last visit at month 24 will be requested to complete an Early Termination visit.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in COPD Assessment Test (CAT) Score | Baseline up to 12 months
  The COPD Assessment Test (CAT) is a questionnaire to assess the health status and quality of life of people with COPD. The questionnaire consists of eight simple statements, which participants answer using a numerical scale. The CAT score ranges from 0 to 40, with lower scores indicating a better health status.

SECONDARY OUTCOMES:
Change from Baseline in CAT Score | Baseline to up to 6 months and 24 months
  The COPD Assessment Test (CAT) is a questionnaire to assess the health status and quality of life of people with COPD. The questionnaire consists of eight simple statements, which participants answer using a numerical scale. The CAT score ranges from 0 to 40, with lower scores indicating a better health status.
Analysis of Socio-demographics, Medical Disease and Treatment History | Baseline
  Demographic data (age, sex [f/m], ethnicity, height, weight, BMI, vaccination status, smoking status, pack years) will be collected.
Analysis of Clinical Disease Characteristics including Exacerbations | Baseline
  Number and severity grade of exacerbations in the year before study start will be assessed.
Analysis of Clinical Disease Characteristics including Lung Function Parameters | Baseline
  Lung function parameters such as forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), FEV1/FVC, total lung capacity (TLC), residual volume (RV), sRtot, Diffusing capacity of the lungs for carbon monoxide (DLCO), DLCO/VA, Rtot, oxygen saturation in the blood will be assessed.
Analysis of Clinical Disease Characteristics including Eosinophils [EOS] Levels | Baseline
  Analysis of clinical disease characteristics including EOS levels.
Analysis of Clinical Disease Characteristics including Fractional Exhaled Nitric Oxide [FeNO] Levels | Baseline
  Analysis of clinical disease characteristics including FeNO levels.
Analysis of Clinical Disease Characteristics including Immunoglobulin E [IgE] Levels | Baseline
  Analysis of clinical disease characteristics including IgE levels.
Analysis of Clinical Disease Characteristics including Current Global Initiative for Chronic Obstructive Lung Disease (GOLD) Grade and Group | Baseline
  Analysis of clinical disease characteristics including current GOLD grade and group.
Analysis of Clinical Disease Characteristics including Smoking Status and Pack Years | Baseline
  Analysis of clinical disease characteristics including smoking status and pack years.
Analysis of Clinical Disease Characteristics including Comorbidities | Baseline
  Current and previous comorbidities (such as chronic rhinosinusitis, asthma, allergies, or cardiovascular comorbidities) will be assessed.
Analysis of Clinical Disease Characteristics including Date of COPD Diagnosis and GOLD Grade/Group at COPD Diagnosis | Baseline
  Analysis of clinical disease characteristics including date of COPD diagnosis and GOLD grade/group at COPD diagnosis.
Annualized Rate of Moderate and Severe COPD Exacerbations | Baseline to up to 12 and 24 months
  Annualized rate of moderate and severe COPD exacerbations after 12 and 24 months versus the year before baseline.
Change in Rate of Moderate and Severe Exacerbations | Baseline to up to 6, 12 and 24 months
  Change in rate of moderate and severe exacerbations will be assessed.
Time to First Moderate or Severe Exacerbation Since Study Start | Baseline to up to 6, 12 and 24 months
  Time to first moderate or severe exacerbation since study start.
Cumulative Moderate and Severe Exacerbations Over Time | Baseline to up to 6, 12 and 24 months
  Cumulative moderate and severe exacerbations over time
Change Over Time in Pre- and Post-Bronchodilator Forced Expiratory Volume in 1 Second (FEV1) | Baseline to up to 6, 12 and 24 months
  Change over time in pre- and post-bronchodilator FEV1 from study start.
Change Over Time in Bronchodilator FEV1/Forced Vital Capacity (FVC) | Baseline to up to 6, 12 and 24 months
  Change over time in pre- and post- bronchodilator FEV1/FVC from study start.
Change Over Time in Modified Medical Research Council (mMRC) | Baseline to up to 6, 12 and 24 months
  Change over time in mMRC from study start.
Number of Missed Workdays due to COPD | Baseline to up to 6, 12 and 24 months
  Number of missed workdays due to COPD during the last year before baseline and after dupilumab treatment.
Number of Hospitalization After Dupilumab Treatment | Baseline to up to 6, 12 and 24 months
  Number of hospitalizations after dupilumab treatment versus the year before study start.
Reason(s) for Initiation of Dupilumab Treatment | Baseline
  Reason(s) for initiation of dupilumab treatment will be evaluated.
Frequency of Adverse Events (AEs) During the Observation Period | Baseline to up to 24 months
  Frequency of AEs will be evaluated during the observation period.
Type of AEs | Baseline to up to 24 months
  Type of AEs will be evaluated during the observation period.
Frequency of Possible Dupilumab-Related Treatment Emergent AEs (TEAEs) | Baseline to up to 24 months
  Frequency of possible dupilumab-related TEAEs will be evaluated during the observational period.
Type of Possible Dupilumab-Related TEAEs | Baseline to up to 24 months
  Type of possible dupilumab-related TEAEs will be evaluated during the observational period.
Occurrence of Product Technical Complaints (PTCs) | Baseline to up to 6, 12 and 24 months
  Occurrence of PTCs will be evaluated.

CONTACTS AND LOCATIONS:
Locations (18):
- Germany (18):
  - Investigational Site Number: DE18, Auerbach
  - Investigational Site Number: DE21, Augsburg
  - Investigational Site Number: DE13, Bad Homburg
  - Investigational Site Number: DE19, Berlin
  - Investigational Site Number: DE02, Berlin
  - Investigational Site Number: DE29, Burgwedel
  - Investigational Site Number: DE01, Darmstadt
  - Investigational Site Number: DE09, Erkelenz
  - Investigational Site Number: DE06, Flensburg
  - Investigational Site Number: DE08, Fürstenwalde
  - Investigational Site Number: DE03, Hamburg
  - Investigational Site Number: DE04, Hamburg
  - Investigational Site Number: DE07, Hohenstein-Ernstthal
  - Investigational Site Number: DE10, Itzehoe
  - Investigational Site Number: DE24, Kaiserslauten
  - Investigational Site Number: DE25, Lüneburg
  - Investigational Site Number: DE20, Marburg
  - Investigational Site Number: DE14, Markkleeberg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org